CLINICAL TRIAL: NCT01366248
Title: Breast Cancer Integrative Oncology: Prospective Matched Controlled Outcomes Study
Brief Title: Integrative Oncology Outcomes Study in Breast Cancer
Acronym: IO-OS-BC
Status: Completed | Type: Observational
Sponsor: Bastyr University (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 09E-1237-01; 1R01AT005873 (NIH)
Record Dates: First submitted 2011-05-31; First posted 2011-06-06 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IO Clinic Breast Cancer Patients: Includes patients who are receiving care for their breast cancer at participating Seattle area IO clinics.
- CSS Match-Control Patients: For each IO clinic patient, an average of two (up to four) matched comparison cases will be recruited from the Washington State Cancer Surveillance System (CSS). Matched comparison cases from CSS will be identified by CSS and confirmed by the FHCRC investigator.

SUMMARY:
This NIH-NCCAM funded epidemiologic research is being conducted as an observational prospective case-control study of the use of Complementary and Alternative Medicine (CAM) and Integrated Oncology (IO) and their effects on breast cancer patients in community settings.

Hypothesis: IO services improve patients' quality of life and decrease cancer recurrence rates in breast cancer patients as compared to women with similar disease states and prognoses who do not receive IO care, and may or may not use CAM treatment on their own.

ELIGIBILITY:
The patients enrolled into the study will include patients who meet the following criteria:

Cohort 1: IO clinic breast cancer patients

1. Confirmed breast cancer of primary breast cancer with ICD9 code of 174.x, 233.0 or V10.3
2. Female
3. ≥18 years of age
4. Can provide signed informed consent
5. 1st IO clinic visit ≤3 months prior to enrollment
6. Can read and understand the questionnaires

Cohort 1A: Sub-cohort of IO clinic patients (cases) who meet the following additional criteria and for whom matched controls have been found from the CSS database.

1. ICD9 code of 174.x or 233.0
2. Primary ductal or lobular breast cancer diagnosis ≤2 years prior to 1st IO clinic visit
3. Minimum of two IO clinic visits within 7 months
4. Provided Baseline Questionnaire

Cohort 2: Matched controls from CSS database for Cohort 1A patients

1. Confirmed breast cancer
2. Female
3. ≥ 18 years of age
4. Can provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants for the study will include patients who are receiving care for their cancer at participating Seattle area IO clinics. An average of two (up to four) matched comparison controls will be recruited from the Washington State CSS.
  All breast cancer patients seeking care at the participating IO clinics who meet inclusion/exclusion criteria are eligible to participate in this study. Matched comparison cases from CSS will be identified by CSS and confirmed by the FHCRC investigator.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2010-08; Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Aim 1: Describe treatments received by breast cancer patients receiving physician level practitioner IO care and the cost of IO care. | Baseline, 6, 12, 24, 36, 48, and 60 months post study enrollment.
  Will also describe how long after diagnosis women with breast cancer seek IO care and differences in IO care prescriptions associated with when, in a woman's course of treatment, she seeks care. This patient cohort will consist of all female patients with breast cancer seeking IO clinic care. Our analyses will describe how long after diagnosis women with breast cancer seek IO care and describe differences in IO care prescriptions associated with when, in a woman's course of treatment, she seeks care.
Aim 2: Compare health-related quality of life (HRQOL) experienced by a group of breast cancer patients receiving IO care with HRQOL of a group of matched comparison women. | 6-60 months post-enrollment
  Comparison will be between breast cancer patients living in the same geographic area with similar prognostic characteristics (age, stage of cancer at diagnosis, estrogen receptor/ progesterone receptor (ER/PR) status, race, ethnicity, and marital status) at the time of their initial diagnosis with breast cancer who did not receive IO care. We will identify an average of three (up to four each) matched controls for each eligible IO clinic cancer patient from the Western Washington CSS database and to invite them to enroll in the outcomes study.

SECONDARY OUTCOMES:
Aim 3: Collect pilot data on survival, comorbidities, and abnormal laboratory values. | 6-60 months post-enrollment
  Collect pilot data on disease-free, progression free, and overall survival, as well as comorbidities and abnormal laboratory values at 6 months post-enrollment for all Cohort 1 and Cohort 2. We will collect data at 1 year post-enrollment and then yearly on disease-free, progression free, and overall survival, as well as comorbidities for as long as funding is available in a nested cohort of IO breast cancer patients (Cohort 1A) and their matched comparison group who did not receive care at any of the IO clinical sites (Cohort 2).
Aim 4: Describe and compare CAM treatments | Baseline, 6, 12, 24, 48, and 60 months
  Describe and compare the frequency of use of a variety of CAM treatments used by breast cancer patients who do (Cohort 1A) and do not (Cohorts 2A and 2B) receive IO care from an IO specialist.
Aim 5: Compare the HRQOL of women who self-prescribe CAM with those who do not | Baseline and 6, 12, 24, 36, 48 and 60 months post-enrollment
  To compare baseline and changes in HRQOL in breast cancer patients who self-prescribe CAM (Cohort 2B) matched with comparison women who do not use CAM (Cohort 2A).

CONTACTS AND LOCATIONS:
Overall Officials: Leanna J. Standish, ND, PhD, FABNO, Principal Investigator — Bastyr University; M. Robyn Andersen, PhD, MPH, Principal Investigator — Fred Hutchinson Cancer Center
Locations (6):
- United States (6):
  - Red Cedar Wellness Center, Bellevue, Washington
  - Bastyr Integrative Oncology Research Center, Kenmore, Washington
  - Seattle Integrative Oncology at Providence Integrative Cancer Care, Lacey, Washington
  - Seattle Cancer Treatment & Wellness Center, Renton, Washington
  - Seattle Integrative Oncology at Institute of Complementary Medicine, Seattle, Washington
  - Tree of Health Integrative Medicine, Woodinville, Washington

REFERENCES:
- [Derived] Standish LJ, Dowd F, Sweet E, Dale L, Andersen MR. Do Women With Breast Cancer Who Choose Adjunctive Integrative Oncology Care Receive Different Standard Oncologic Treatment? Integr Cancer Ther. 2018 Sep;17(3):874-884. doi: 10.1177/1534735418769007. Epub 2018 Apr 27. PMID 29701107